CLINICAL TRIAL: NCT03582254
Title: Role of [18F]-FDG Brain PET in Newly Diagnosed Primary Cerebral Lymphoma, in Immunocompetent Patient Older Than 60 Years
Acronym: LOCALYSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOR14101; 2014-002597-37 (EudraCT Number)
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Primary Central Nervous System Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]-FDG PET/MR (Experimental): [18F]-FDG PET/MR will be performed in the Department of Nuclear Medicine - Pitié-Salpêtrière Hospital
  Interventions: Radiation: [18F]-FDG PET/MR

INTERVENTIONS:
Radiation: [18F]-FDG PET/MR — [18F]-FDG PET/MR will be performed in the Department of Nuclear Medicine - Pitié-Salpêtrière Hospital:
  * prior to initiation of chemotherapy (rituximab, methotrexate, procarbazine, vincristine and cytarabine) (PET#1),
  * after two chemotherapy cycles (PET#2),
  * at the end of the first-line chemotherapy regimens (PET#3).

SUMMARY:
Patients older than 60 years account for half of cases of Primary Central Nervous System Lymphoma (PCNSL) and have a poorer outcome. No prognostic or predictive factors exist for survival after initial remission. 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose - Positron Emission Tomography ([18F]FDG-PET) plays a key role in grading and therapy monitoring of systemic diffuse large B-cell type.

LOCALYZE is an ancillary Positron Emission Tomography / Magnetic Resonance (PET/MR) clinical study from BLOCAGE 01 (Pr Hoang-Xuan). The aim is to evaluate the usefulness of [18F]FDG-PET to monitor treatment response in PCNSL older than 60 years (n=56), in complement to multiparametric Magnetic Resonance Imaging (MRI).

Hypothesis The investigators assume that the development of new imaging biomarker extracted from PET imaging and multiparametric MRI, could improve the assessment of treatment response in PCNSL.

DETAILED DESCRIPTION:
[18F]-FDG PET/MR will be performed in the Department of Nuclear Medicine - Pitié-Salpêtrière Hospital:

* prior to initiation of chemotherapy (rituximab, methotrexate, procarbazine, vincristine and cytarabine) (PET#1),
* after two chemotherapy cycles (PET#2),
* at the end of the first-line chemotherapy regimens (PET#3).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed primary cerebral lymphoma
* Age ≥60 years
* Pathology proven diagnosis or positive cytology of the Cerebrospinal Fluid (CSF) or vitreous
* Karnofsky Performance Status ≥40
* No evidence of systemic Non-Hodgkin lymphomas (NHL) (body CT scan, bone marrow biopsy)
* Adequate haematological, renal and hepatic function
* Calculated creatinine clearance > 40 ml/min

Exclusion Criteria:

* Uncontrolled diabetes with fasting glycaemia > 200 mg/dL
* Sensitivity to active substance in [18F]-FDG
* Calculated creatinine clearance < 40 ml/min
* No contraindication to MRI (magnetic resonance imaging)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival calculated from the date of completion of the end of chemotherapy PET | 6 months
  To evaluate the predictive value of [18F]FDG-PET assessment performed at the end-of-treatment (high-dose methotrexate based polychemotherapy), on progression free survival in newly diagnosed PCNSL with age ≥60 years (n=56).

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rozenblum L, Houillier C, Baptiste A, Soussain C, Edeline V, Naggara P, Soret M, Causse-Lemercier V, Willems L, Choquet S, Ursu R, Galanaud D, Belin L, Hoang-Xuan K, Kas A. Interim FDG-PET improves treatment failure prediction in primary central nervous system lymphoma: An LOC network prospective multicentric study. Neuro Oncol. 2024 Jul 5;26(7):1292-1301. doi: 10.1093/neuonc/noae029. PMID 38366824